CLINICAL TRIAL: NCT02299011
Title: Comparison of Biomatrix and Orsiro Drug Eluting Stent in Angiographic Result in Patients With All-comer Patients With Coronary Artery Disease : A Multicenter, Randomized, Open Label Study (BIODEGRADE Study)
Brief Title: Comparison of Biomatrix and Orsiro Drug Eluting Stent
Acronym: BIODEGRADE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: Wonju Severance Christian Hospital (Other); Korea University Guro Hospital (Other); Gangnam Severance Hospital (Other); Chungnam National University Hospital (Other); The Catholic University of Korea (Other); Korea University Anam Hospital (Other); Kosin University Gospel Hospital (Other); KangWon National University Hospital (Other); Gachon University Gil Medical Center (Other)
Responsible Party: Principal Investigator, Chang-Hwan Yoon, Assistant professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B1403-244-002
Record Dates: First submitted 2014-11-17; First posted 2014-11-24 (Estimated); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Coronary Artery Disease; Myocardial Ischemia
Keywords: Biomatrix drug eluting stent; Orsiro drug eluting stent; Coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia | interventions — Biosensing Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Orsiro drug eluting stent (Experimental): Orsiro drug eluting stent
  Interventions: Device: Orsiro drug eluting stent
- Biomatrix drug eluting stent (Active Comparator): Biomatrix drug eluting stent
  Interventions: Drug: Biomatrix drug eluting stent

INTERVENTIONS:
Device: Orsiro drug eluting stent — Orsiro Hybrid drug eluting stent
  Other Names: Orsiro drug eluting stent (Biotronik AG, Bulach, Switzeland)
  Arms: Orsiro drug eluting stent
Drug: Biomatrix drug eluting stent — Biomatrix Flex drug eluting stent
  Other Names: Biomatrix drug eluting stent (Biosensors,Newport Beach,USA)
  Arms: Biomatrix drug eluting stent

SUMMARY:
The primary objective of the BIODEGRADE study is to evaluate clinical efficacy of the Orsiro drug-eluting stent compared with Biomatrix drug-eluting stent, both of which have biodegradable polymer for the treatment of all-comers' coronary artery diseases.

DETAILED DESCRIPTION:
The rate of in-stent restenosis after percutaneous coronary intervention (PCI) has decreased since the launching of drug-eluting stents (DES). However, restenosis still remains a problem since PCI is being performed on more complex, calcified, tortuous and tough lesions. Furthermore, there is still a controversy on whether these DES are more thrombogenic than bare metal stent (BMS) because of inflammation related to the polymer coating and delayed vessel healing due to the eluted drug despite of reduced restenosis. Therefore, works aiming to reduce both restenosis and thrombotic event are still on-going in the field of interventional cardiology, and there has been a rush of various third generation DES with "biodegradable polymer". Recently, Orsiro hybrid DES (Biotronik AG, Bulach, Switzeland) has been developed. The Orsiro DES incorporated optimally combined two kind of polymer onto thinner cobalt-chromium backbone (60um) compared with earlier type of DES. The BIOlute® active component is a bioabsorbable polymer matrix combined with an anti-proliferative drug, sirolimus, that is released in a controlled manner leaving only the PROBIO® coated stent in the long-term. The PROBIO® passive coating encapsulates the stent and eliminates interaction between the metal stent and the surrounding tissue. To date, Orsiro stent showed excellent results in terms of late lumen loss at 9 months in first-in-man single arm trial comparing the historical results of other DES (BIOFLOW-I trial), and RCT with non-inferiority design, comparing late lumen loss at 9 months of Orsiro versus everolimus-eluting stent (Xience prime®) is ongoing (BIOFLOW-II trial). However, there have been no trials comparing the Orsiro stent versus the Biomatrix stent (Biosensors Inc, Newport Beach, CA, USA).

This multicenter, randomized, open label, parallel arm study will evaluate whether the innovative newer generation stent, Orsiro hybrid DES, is non-inferior to the third generation stent, Biomatrix stent, in terms of 18 months late lumen loss.

ELIGIBILITY:
Inclusion Criteria:

1. General Inclusion Criteria

   1. Subject must be at least 18 years of age.
   2. Subject is able to verbally confirm understandings of risks, benefits and treatment alternatives of receiving the Biomatrix flex stents or Orsiro stents, and he/she or his/her legally authorized representative provides written informed consent prior to any study related procedure.
   3. Subject must have significant lesion (>50% by visual estimate) in any of the coronary arteries, venous or arterial bypass grafts.
   4. Subject must have evidence of myocardial ischemia (e.g., stable, unstable angina, recent infarction, silent ischemia, positive functional study or a reversible changes in the electrocardiogram (ECG) consistent with ischemia). In subjects with diameter stenosis > 70%, evidence of myocardial ischemia does not have to be documented.
2. Angiographic Inclusion Criteria

   1. Target lesion(s) must be located in coronary artery, venous or arterial bypass graft with diameter of ≥ 2.5 mm and ≤ 4.5 mm.
   2. Target lesion(s) must be amenable for percutaneous coronary intervention.

Exclusion Criteria:

1. The patient has a known hypersensitivity or contraindication to any of the following medications: Heparin, Aspirin, Clopidogrel, Cilostazol, Prasugrel, Ticagrelor, Biolimus, Sirolimus, Contrast media (Patients with documented sensitivity to contrast media which can be effectively premedicated with steroids and diphenhydramine [e.g. rash] may be enrolled. Those with true anaphylaxis to prior contrast media, however, should not be enrolled.)
2. Systemic (intravenous) Biolimus or Sirolimus use within 12 months.
3. Female of childbearing potential, unless a recent pregnancy test is negative, who possibly plan to become pregnant any time after enrollment into this study.
4. History of bleeding diathesis, known coagulopathy (including heparin- induced thrombocytopenia), abnormal hemogram (Hb<10g/dL or PLT count <100,000/μL) or will refuse blood transfusions
5. Patients with severe LV systolic dysfunction (LVEF<25%) or cardiogenic shock
6. Gastrointestinal or genitourinary bleeding within the prior 2 months, or major surgery within 2 months.
7. Non-cardiac co-morbid conditions are present with life expectancy <1 year or that may result in protocol non-compliance (per site investigator's medical judgment).
8. Patients who are actively participating in another drug or device investigational study, which have not completed the primary endpoint follow- up period.
9. Symptomatic heart failure

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2341 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Target lesion failure (TLF) | 18 months
  TLF is a composite of cardiac death, target vessel-related myocardial infarction and ischemia-driven target lesion revascularization as measured by percent of participants with adverse events

SECONDARY OUTCOMES:
All death | 18 months
  All-cause death as measured by percent of participants with adverse events
All death | 36 months
  All-cause death as measured by percent of participants with adverse events
Cardiac death | 18 months
  cardiac death as measured by percent of participants with adverse events
Cardiac death | 36 months
  cardiac death as measured by percent of participants with adverse events
Target vessel-related MI and all MI | 18 months
  Target vessel-related MI and all MI as measured by percent of participants with adverse events subdivided as q wave and non-q wave
Target vessel-related MI and all MI | 36 months
  Target vessel-related MI and all MI as measured by percent of participants with adverse events subdivided as q wave and non-q wave
Stent thrombosis | 18 months
  Stent thrombosis (definite/possible/probable) as measured by percent of participants with adverse events
Stent thrombosis | 36 months
  Stent thrombosis (definite/possible/probable) as measured by percent of participants with adverse events
Net clinical outcome including bleeding (major and minor) as measured by percent | 18 months
  Net clinical outcome including bleeding (major and minor) as measured by percent of participants with adverse events
Net clinical outcome including bleeding (major and minor) as measured by percent | 36 months
  Net clinical outcome including bleeding (major and minor) as measured by percent of participants with adverse events
In-stent & In-segment late loss | 18 months
  In-stent & In-segment late loss as measure by post-PCI and F/U QCA
In-stent & In-segment late loss | 36 months
  In-stent & In-segment late loss as measure by post-PCI and F/U QCA
In-stent & In-segment % diameter stenosis | 18 months
  In-stent & In-segment % diameter stenosis as measure by post-PCI and F/U QCA
In-stent & In-segment % diameter stenosis | 36 months
  In-stent & In-segment % diameter stenosis as measure by post-PCI and F/U QCA
Degree of stent strut endothelialization and malapposition on OCT | 18 months
  Degree of stent strut endothelialization and malapposition on OCT as measure by post-PCI and F/U OCT analysis
Degree of stent strut endothelialization and malapposition on OCT | 36 months
  Degree of stent strut endothelialization and malapposition on OCT as measure by post-PCI and F/U OCT analysis
Target lesion failure (TLF) | 36 months
  TLF is a composite of cardiac death, target vessel-related myocardial infarction and ischemia-driven target lesion revascularization as measured by percent of participants with adverse events

CONTACTS AND LOCATIONS:
Overall Officials: In-Ho Chae, MD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National Universtiy Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

REFERENCES:
- [Background] Hamon M, Niculescu R, Deleanu D, Dorobantu M, Weissman NJ, Waksman R. Clinical and angiographic experience with a third-generation drug-eluting Orsiro stent in the treatment of single de novo coronary artery lesions (BIOFLOW-I): a prospective, first-in-man study. EuroIntervention. 2013 Jan 22;8(9):1006-11. doi: 10.4244/EIJV8I9A155. PMID 23339805
- [Derived] Kwun JS, Park JJ, Kang SH, Kim SH, Yoon CH, Suh JW, Youn TJ, Cha KS, Lee SH, Hong BK, Rha SW, Kang WC, Chae IH. Interpreting clinical outcomes using different strut thickness in coronary artery disease: insights from vascular imaging analysis. Front Cardiovasc Med. 2025 Mar 4;12:1491607. doi: 10.3389/fcvm.2025.1491607. eCollection 2025. PMID 40104139
- [Derived] Yoon CH, Kwun JS, Choi YJ, Park JJ, Kang SH, Kim SH, Suh JW, Youn TJ, Kim MK, Cha KS, Lee SH, Hong BK, Rha SW, Kang WC, Lee JH, Kim SH, Chae IH. BioMatrix Versus Orsiro Stents for Coronary Artery Disease: A Multicenter, Randomized, Open-Label Study. Circ Cardiovasc Interv. 2023 Jan;16(1):e012307. doi: 10.1161/CIRCINTERVENTIONS.122.012307. Epub 2022 Dec 7. PMID 36475473